CLINICAL TRIAL: NCT02552056
Title: The Effect of Integrating Child and Adolescent Mental Health Into Primary Health Care and Traditional Healers' Practice: a Randomized Controlled Trial in Eastern Uganda
Brief Title: The Effect of Integrating CAMH Into PHC and Traditional Healers' Practice in Uganda: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Principal Investigator, Angela Akol, PhD candidate, University of Bergen
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HS 1874
Record Dates: First submitted 2015-09-14; First posted 2015-09-16 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Community Mental Health Services
Keywords: Child Adolescent Mental Integration PHC Traditional Healers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAMH training (Experimental): Intervention clinics will receive a CAMH integration package comprising of:
  * Training PHC workers (midwives, nurses and/or clinical officers) on how to screen and refer for CAMH, based on WHO mhGAP implementation guide.
  * Support supervision in the clinics to reinforce training and provide on-job support to PHC staff.
  * Provision of job aids and training materials
  Interventions: Other: CAMH training
- No CAMH training (No Intervention): Clinics will continue to provide the standard of care.

INTERVENTIONS:
Other: CAMH training — Training of PHC workers included in the study for 5 days to screen children and adolescents for CAMH conditions, based in the mhGAP curriculum for non-specialist health providers.
  Arms: CAMH training

SUMMARY:
This randomized controlled trial will compare the effect of a CAMH integration package on yield of CAMH cases compared to non-CAMH integrated sites. It will be conducted among nurses, midwives and clinical officers who provide PHC services to children and adolescents in 42 health centers; and eligible traditional healers.

DETAILED DESCRIPTION:
The overall goal of the study is to increase access to mental health services for children and adolescents in Uganda by improving entry through primary health care workers and traditional healers.

The main objective of the study is to measure the effect of integrating child and adolescent mental health (CAMH) into primary health care (PHC) and into traditional healers' services on CAMH case identification in 2 districts in Eastern Uganda, so as to improve entry into mental health services.

The specific objectives are:

1. To estimate the effect of CAMH integration into PHC on case identification, measured by the number of new non- epilepsy CAMH diagnoses.
2. To assess the feasibility and effect of integrating CAMH into traditional healers practice, measured by the number of CAMH referrals from community to clinics per month.
3. To assess the acceptability of CAMH integration among PHC workers and traditional healers
4. To estimate the costs associated with the integration of CAMH into PHC and traditional medicine

ELIGIBILITY:
Inclusion Criteria:

* 1. Public (government health system) 2. No psychiatric nurse allocated

Exclusion Criteria:

* mhGAP training in the previous 3 years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Proportion of clinics which recorded at least one non-epilepsy CAMH diagnosis in the intervention compared to the control group. | 3 months

OTHER OUTCOMES:
Change in CAMH knowledge pre-and post-training | 5 days

REFERENCES:
- [Derived] Akol A, Makumbi F, Babirye JN, Nalugya JS, Nshemereirwe S, Engebretsen IMS. Does mhGAP training of primary health care providers improve the identification of child- and adolescent mental, neurological or substance use disorders? Results from a randomized controlled trial in Uganda. Glob Ment Health (Camb). 2018 Sep 10;5:e29. doi: 10.1017/gmh.2018.18. eCollection 2018. PMID 30455964